CLINICAL TRIAL: NCT05170685
Title: Expanded Access for Fixed-Dose Combination of Nivolumab Plus Relatlimab
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA224-129
Record Dates: First submitted 2021-11-17; First posted 2021-12-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Nivolumab plus Relatlimab FDC

SUMMARY:
This is an expanded access designed to provide access to fixed-dose combination of nivolumab plus relatlimab for eligible participants.

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Pre-approval Access (PAA) Healthcare Practitioner Requests — https://www.bms.com/healthcare-providers/early-patient-access-to-investigational-medicine/investigational-drugs-available.html
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm